CLINICAL TRIAL: NCT03384901
Title: The Results of Pars Plana Vitrectomy in Diabetic Macular Edema
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0109-17-HYMC
Record Dates: First submitted 2017-12-20; First posted 2017-12-28 (Actual); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Vitrectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: vitrectomy — Pars plana vitrectomy and ILM (internal limiting membrane) peeling

SUMMARY:
This study will be a retrospective analysis of vitrectomy results in patients suffering from diabetic macular edema.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic macular edema patients after vitrectomy

Exclusion Criteria:

* All others

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending the Hillel Yaffe Medical Center Ophthalmology Clinic
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | 6 months
  Visual acuity will be measured using the Snellen Chart before and after vitrectomy

SECONDARY OUTCOMES:
Macular thickness | 6 months
  Macular thickness will be measured using Optical Coherence Tomography before and after vitrectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Hille Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No